CLINICAL TRIAL: NCT03406559
Title: Comparison of TMJ Disc-condyle-fossa Relationship, After Fixed Orthodontic Treatment of Adolescent Males With Skeletal Class II, Angle's Class II Division 2 Malocclusion Treated Initially With Removable Functional Appliance: an MRI Study.
Brief Title: TMJ Adaptations by Orthodontic Treatment in Adolescent Males With Angle's Class II Division 2 Malocclusion: MRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: deepak sindhu
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Class II Division 2 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Orthodontics

STUDY DESIGN:
Intervention Model Description: study on 14 male adolescent patients having skeletal class II, Angle's class II division 2 malocclusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- orthodontic treatment (Other): fixed orthodontic treatment in adolescent males initially treated with removable functional appliances for skeletal class II, Angle's class II division 2 malocclusion.
  Interventions: Other: orthodontic treatment

INTERVENTIONS:
Other: orthodontic treatment — fixed orthodontic treatment in adolescent males initially treated with removable functional appliances for skeletal class II, Angle's class II division 2 malocclusion,
  Other Names: fixed mechanotherapy

SUMMARY:
the aim of this study is to document the changes brought about in the internal anatomic relationships of the TMJ complex , positional changes of glenoid fossa with respect to adjacent cranial structures after completion of fixed orthodontic treatment in adolescent males initially treated with removable functional appliances for skeletal class II, Angle's class II division 2 malocclusion

DETAILED DESCRIPTION:
Angle's class II division 2 malocclusion is subtype of Angle's class II malocclusion with unique facial, dental and craniofacial features which differentiate it from other malocclusions so much that it has been said to be a syndrome itself. Its frequency lies between 1.5 and 5% of all malocclusions found in a white western population.. Condyle position changes from anterior to posterior with age in class II division 2 cases. The use of functional orthopedic appliances to correct Class II malocclusions associated with retrognathic mandibles is indicated for the first phase of orthodontic treatment. A second phase of treatment is undertaken with fixed orthodontic appliances to obtain occlusal refinement. Although various investigations have shown the efficiency of this method of treatment, the mechanism by which the temporomandibular joint (TMJ) responds to the treatment is controversial.

Various techniques have been used to image the TMJ which include Magnetic Resonance Imaging (MRI), Cephalograms, Orthopantomograms , Tomograms , Bone scintigraphy with radiologic markers like 99mTc-MDP, Arthroscopy and Arthrography , CT scanning, Cone Beam Computed Tomography (CBCT).

Magnetic Resonance Imaging (MRI), a multiplanar imaging technique, has the advantage of giving an accurate assessment of both the bony and the soft tissues. This technique is believed to be non-invasive, radiation free and gives more superior contrast resolution than any other imaging modality. MRI is considered the imaging modality of choice for assessment of internal derangements of the temporomandibular joint. Bony structures and especially soft tissues of the TMJ can be examined by means of MRI and the relations of the tissues with each other can be evaluated.

MRI studies have been done on fixed functional appliances which show significant displacement of condyle during treatment but later condyles returned to pre treatment positions at the end of fixed functional appliance treatment. Results documented in fixed functional appliance may not be same in removable appliances. Effects of removable functional appliances on the condyle-glenoid fossa (C-GF) complex have been studied with respect to the Frankel, Activator, Twin block and Bionator appliances.It should be noted that all of above studies are limited to the phase of removable functional appliance therapy only in Class II division 1 and no MRI study has attempted to evaluate the changes in the position of the Condyle-Glenoid Fossa (C-GF) complex treated with removable functional appliance therapy, followed by fixed orthodontic treatment in Class II division 2 malocclusion.

No studies have been done on bi-phasic treatment of skeletal class II, Angle's class II division 2 involving removable functional appliances in the first phase followed by fixed orthodontic treatment in second phase.

Therefore, the aim of this study is to document the changes brought about in the internal anatomic relationships of the TMJ complex , positional changes of glenoid fossa with respect to adjacent cranial structures after completion of fixed orthodontic treatment in adolescent males initially treated with removable functional appliances for skeletal class II, Angle's class II division 2 malocclusion,

MATERIALS AND METHODS

It is a longitudinal clinical trial to evaluate TMJ disc-condyle-fossa relationship using MRI scan following bi-phasic therapy in skeletal Class II, Angle's class II division 2 malocclusion in adolescent males.

The present study will be conducted in the Department of Orthodontics and Dentofacial Orthopedics, PGIDS, in association with the Department of Radiology, PGIMS, and Department of Oral Radiology, PGIDS, Pt B. D. Sharma University of Health Sciences, Rohtak.

Ethical clearance- The study will be carried out in humans after the institutional approval obtained from ethical committee.

Source of Data The study sample will consist of the subjects from the Department of Orthodontics and Dentofacial Orthopedics, PGIDS , who will be successfully completing the prefunctional and functional appliance therapy for correction of skeletal class II, Angle's class II division 2 malocclusion and will be ready for fixed orthodontic treatment for final finishing and detailing of occlusion

INFORMED CONSENT OF THE PATIENT

A valid, bilingual informed written consent of the patient or parent/guardian will be obtained from the patient before registering the patient in this clinical study. Patients will be informed of all the theoretical risks and benefits of the interventions under test.

Intervention and design of study The study sample will consist of those 14 adolescent males who had been treated initially with pre functional and functional appliance therapy for skeletal Class II, Angle's class II division 2 malocclusion and had following MRI scans done during the treatment

1. Stage- A (pre-treatment),
2. Stage- B (after pre-functional therapy)
3. Stage- C (After completion of Functional Appliance Therapy) These patients will be further treated with fixed orthodontic treatment for final finishing and detailing and an MRI will be taken after debonding of fixed orthodontic appliance (stage D). MRI scans thus obtained will be evaluated for documenting changes in the morphology and anatomic positions of condylar head, articular disc and glenoid fossa and will be traced for the various angular and linear metric measurements MRI scans of the TMJ will be obtained with a 1.5 Tesla Philips Intera Nova Gradient (Netherlands) scanner equipped with Sense Head 6 channel coil for simultaneous imaging of right and left joints. Sagittal images will be taken perpendicular to the long axis of the condylar head and the coronal images will be taken parallel to the long axis of the condylar head. The images will be recorded in maximum intercuspation after debonding of fixed orthodontic appliance. The MRI protocol will include PD TSE (Turbo Spin Echo) sequence (TR 1500/ TE 30/ FoV 150x150 mm) T1 spin echo sequences (TR 450⁄TE 15⁄FoV 160x160 mm) and T2 TSE sequence (TR 2424⁄ TE 100⁄FoV 160x160 mm).

FIXED MECHANOTHERAPY TREATMENT PHASE

The sample will be having cases in class I/ superclass I molar relation and lateral open bite may be present in premolar regions after the completion of functional phase. The final fixed orthodontic phase will be taken up for the final finishing and detailing of the occlusion after the retentive phase of functional appliance therapy is completed. It involves banding and bonding of both upper and lower arches with MBT 0.022" appliance. Progressive wire sequences to be used are 0.014" NiTi, 0.016" NiTi, 0.018" NiTi, 0.017" x 0.025" NiTi, 0.019"x 0.025" NiTi, , 0.019"x 0.025" S.S., 0.014" S.S. Once stainless steel archwires are in place, class II elastics may be prescribed to the patient to prevent relapse of class I molar relation achieved. Cases are to be finished in class I molar intercuspation with normal overjet and overbite. Appliance will be debonded and final MRI (stage D) will taken for all the patients. Hawley's retainer with anterior bite plane will serve for retention of achieved results

Evaluation of MRI stages This will be done with the help of various angular and linear measurements like the eminence angle, the sagittal disc position measured in relation to two reference lines: the posterior condylar line (PC line) and the Frankfurt Horizontal plane (FH Plane), the coronal disc position , Sagittal condylar concentricity 5) The glenoid fossa angle, Condyle and glenoid fossa displacements and Superior joint space

Statistical analysis The final data recorded will be processed by standard statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Cases with moderate skeletal Class II bases with mandibular retrognathia, Angle's Class II division 2 malocclusion treated initially with prefunctional and functional appliance therapy in their active growth period and will be ready for fixed orthodontic treatment and have had MRI done at following stages:

  1. Stage- A (pre-treatment)
  2. Stage- B (after pre-functional therapy)
  3. Stage-C (After completion of functional appliance therapy)

Exclusion Criteria:

* Patients with any internal derangement or pathology of TMJ.
* History of previous orthodontic interventions or systemic diseases affecting bone metabolism.
* Growth abnormality.
* Bleeding disorders.
* Patients with facial asymmetry.

Ages: 13 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — males
Enrollment: 14 (Actual)
Dates: Start 2016-10-29 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
sagittal condyle concentricity | 12 months
  measured in percentage displacement of condyle in the glenoid fossa
sagittal disc position | 12 months
  measured in degrees from references from Frankfurt Horizontal plane and Posterior Condylar line.
Linear glenoid fossa displacement | 12 months
  measured in millimetres, distance from external auditary meatus to centre of condylar head and Posterior glenoid spine
Superior joint space | 12 months
  measured in millimetres, distance between most superior point on glenoid fossa and superiormost point on condyle
eminence angle | 12 months
  measured in degrees, the angle of anterior slope of glenoid fossa in relation to Frankfurt Horizontal plane and Posterior Condylar line
Glenoid fossa angle | 12 months
  measured in degrees, angle between anterior slope and posterior slope of glenoid fossa
coronal disc position | 12 months
  relative position on the equal tenths on condyle. negative value representing lateral side and positive value indicating the medial side of the disc

CONTACTS AND LOCATIONS:
Overall Officials: deepak sindhu, mds student, Principal Investigator — PGIDS Rohtak, Haryana

IPD SHARING:
Plan to Share IPD: Undecided
the aim of this study is to document the changes brought about in the internal anatomic relationships of the TMJ complex , positional changes of glenoid fossa with respect to adjacent cranial structures after completion of fixed orthodontic treatment in adolescent males initially treated with removable functional appliances for skeletal class II, Angle's class II division 2 malocclusion